CLINICAL TRIAL: NCT00943644
Title: Determination of Sensitivity of a Dual-Headed Small Field of View Gamma Camera for the Detection of Small Breast Lesions
Brief Title: Pre-biopsy With Dynamic Acquisitions
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Michael O'Connor, Ph.D., Mayo Clinic
Other Study IDs: 17-05; BCTR0504394
Record Dates: First submitted 2008-11-10; First posted 2009-07-22 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: MBI; Breast; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Molecular Breast Imaging (MBI) — To determine the sensitivity of MBI
Device: CZT semiconductor detectors — Dual headed CZT semiconductor detectors

SUMMARY:
This study is being done to test the ability of an investigational mammography camera to find small tumors in patients' breasts.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be asked to remove your clothes from the waist up and put on a gown. A female technologist will give you an injection of Tc-99m sestamibi in a vein in your arm. This is a drug routinely used for breast imaging. About 10 minutes after your injection, you will be asked to sit in a chair for about 40 minutes. The technologist will position your breast between two small cameras. The cameras will apply a very light compression to your breast to make sure there is no movement during the picture. We will take two pictures of each breast. Each picture takes 10 minutes. You will also be asked to fill out a short questionnaire. If you are found to have additional breast lesions, your doctor and radiologist will be notified so that additional imaging or biopsies can be performed.

ELIGIBILITY:
Inclusion Criteria:

* Have a lesion on Mammogram, Ultrasound or MRI that measured < 2 cm and considered suspicious or suggestive of malignancy
* Scheduled for biopsy of lesion
* > 18 years of age
* Negative pregnancy test, postmenopausal, or surgically sterilized

Exclusion Criteria:

* Prior needle biopsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are scheduled to have a biopsy at the Mayo Clinic in Rochester, MN and have a lesion less the 2 cm
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2005-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the sensitivity of the dual-head system relative to single-head for detection of sub 10 mm breast lesions, and to determine the number of images that need to be acquired. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael K. O'Connor, Ph.D., Principal Investigator — Mayo Clinic; Deborah J. Rhodes, M.D., Principal Investigator — Mayo Clinic; Douglas A. Collins, M.D., Principal Investigator — Mayo Clinic; Carrie B. Hruska, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States